CLINICAL TRIAL: NCT03331068
Title: Memorial Anxiety Scale for Patients With Prostate Cancer: French Validation, Links With Quality Of Life and Future Temporal Perspective.
Brief Title: French Validation of the Memorial Anxiety Scale for Patients With Prostate Cancer.
Status: Completed | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: MAC-PROSTATE-IPC 2016-009
Record Dates: First submitted 2017-10-02; First posted 2017-11-06 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with prostate cancer: online questionnaire of MAX-PC
  Interventions: Behavioral: online questionnaire of MAX-PC

INTERVENTIONS:
Behavioral: online questionnaire of MAX-PC — Scale measuring of the anxiety specific of prostate cancer, French version.

SUMMARY:
A specific scale allowing the measure of anxiety of patients with protate cancer has been designed and validated but the French version needs to be validated. This study aims at validating the French translation of this scale.

DETAILED DESCRIPTION:
The psychological difficulties encountered by patients with prostate cancer are widely known. There are, however, problems in the identification of certain disorders that require appropriate psychological management. In order to diagnose patients with anxiety more finely, a prostate cancer-specific anxiety measurement scale (MAX-PC) was developed and validated. This scale includes three sub-dimensions: anxiety related to prostate cancer, anxiety related to the PSA assessment and fear of recurrence. This scale generally has good psychometric properties which are found in different populations and in different countries. The dimensions of the MAX-PC correlate with other anxiety measurement scales such as Beck or HADS, but do not show redundancy: it captures a specific anxiety related to the experience of patients with prostate cancer.

To date, this sclae is not validated in French, and its use in the frame of clinical trials or in routine practice require a first validation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prostate cancer diagnosed within 12 months

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists in adult patients with prostate cancer diagnosed within 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Total anxiety score assessed by the Memorial Anxiety Scale for Prostate Cancer (MAX-PC scale) | At inclusion
  The scale is divided in 3 subscales: Prostate cancer Anxiety ; PSA anxiety and Fear of Recurrence. The total score of the scale ranges from 0 to 54, with 54 indicating maximum anxiety. Scores of the Prostate anxiety scale range from 0 to 33 ; with 33 indicating maximum anxiety. Scores of the PSA anxiety scale range from 0 to 9 ; with 9 indicating maximum anxiety. Score of the Fear of Recurrence scale range from 0 to 12; with 12 indicating maximum anxiety. The total score is the sum of the 3 subscales scores.

SECONDARY OUTCOMES:
Quality of Life (QoL) scores assessed by the SF-12 scale | At inclusion
  12-item Short Form Health Survey (SF12), is a multipurpose generic measure oh health status. The SF-12 is weighted and summed to provide easily interpretable scales for physical and mental health.
  Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100 where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. Higher values represent a better outcome.
Anxiety score assessed by the HADS scale | At inclusion
  The scores for anxiety can range from 0 to 21, depending on the presence and severity of the symptom. Patients with a score higher than 7 are detected as having at least mild anxiety.
Depression score assessed by the HADS scale | At inclusion
  The scores for depression can range from 0 to 21, depending on the presence and severity of the symptom. Patients with a score higher than 7 are detected as having at least mild depression.

CONTACTS AND LOCATIONS:
Overall Officials: Gwenaelle GRAVIS, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No